CLINICAL TRIAL: NCT01388517
Title: A Double Blind Randomized Trial, Placebo-controled of 0.0003% Calcitriol Ointment Versus 0.1% Tacrolimus Ointment in the Treatment of Pityriasis Alba
Brief Title: Clinical Trial of 0.0003% Calcitriol, 0.1% Tacrolimus, and Petrolatum for the Treatment of Pityriasis Alba
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad Autonoma de San Luis Potosí (Other)
Collaborators: Hospital Central "Dr. Ignacio Morones Prieto" (Other)
Responsible Party: Principal Investigator, Juan Pablo Castanedo Cazares, Clinical Professor of dermatology, Universidad Autonoma de San Luis Potosí
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PA-CALTAC
Record Dates: First submitted 2011-06-30; First posted 2011-07-06 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: Pityriasis Alba
Keywords: Pityriasis alba; Tacrolimus; Calcitriol; Petrolatum
MeSH Terms: conditions — Dandruff | interventions — Tacrolimus; Calcitriol; Petrolatum

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Calcitriol (Active Comparator): Repigmentation treatment for the relief of hypopigmented pityriasis alba lesions
  Interventions: Drug: Calcitriol
- Tacrolimus (Active Comparator): Treatment for the relief of hypopigmented pityriasis alba lesions
  Interventions: Drug: Tacrolimus
- Petrolatum (Placebo Comparator): Petrolatum treatment for the relief of hypopigmented pityriasis alba lesions
  Interventions: Drug: Petrolatum

INTERVENTIONS:
Drug: Tacrolimus — 0.1% tacrolimus ointment to apply twice a day for 9 weeks on pytiriasis alba plaques.
  Other Names: Protopic; FK506 ointment
  Arms: Tacrolimus
Drug: Calcitriol — 0.0003% calcitriol ointment to apply twice a day for 9 weeks on pytiriasis alba plaques.
  Other Names: Silkis; Topical Vitamin D analogs
  Arms: Calcitriol
Drug: Petrolatum — Petrolatum ointment to apply twice a day for 9 weeks on pytiriasis alba plaques.
  Other Names: Vaseline; Acuaphore
  Arms: Petrolatum

SUMMARY:
Pityriasis alba (PA) is a frequent cause of consultation in tropical areas due to its chronic course, trend to relapse and aesthetic impact. Currently, no treatment is widely accepted. The objective is to assess the calcitriol and tacrolimus ointment efficacy in the treatment of PA compared with petrolatum. Twenty lesions on the face greater than 3 cm, in individuals of phototype IV-V, aged 3-18 years are going to be randomly assigned to receive petrolatum, calcitriol, and tacrolimus twice daily. No photoprotection is going to be indicated, and hygienic habits will not be modified. Patients will be evaluated at baseline and for 9 weeks, by means of Transepidermal Water Loss (TEWL), colorimetry, clinically and by photography control.

DETAILED DESCRIPTION:
Pityriasis alba (PA) is a benign inflammatory dermatosis affecting about 5% of infantile population, frequently seen in tropical areas of the world. This entity has received many synonymous such as chronic impetigo and erythema streptogenes, but its actual name was given from Hazen. PA is also considered a minor criterion for the diagnosis of atopic dermatitis. It is characterized by hypopigmented, irregular plaques with well-defined borders, covered by fine scales; it affects mainly face, limbs and occasionally thorax.

Its etiology is still unknown, although infectious mechanisms and vitamin and minerals deficiencies have been implicated, a causal relationship has not been recognized. However, excessive and unprotected sun exposure is considered the most important causal factor involved. However, studies from stratum corneum from of PA lesions have described defects in hygroscopicity and water-holding capacity detectable by water sorption-desorption test, this suggests that the condition is similar to a dermatitic change and its hypopigmentation may be consequence of a postinflammatory mechanism.

The study population will include at least 20 lesions in individuals with phototype IV-V, affected symmetrically by PA on the face. Their selected age will be less than 18 years. Patients with other dermatoses, including atopic dermatitis, use of any systemic or topical medication during the past 4 weeks will be excluded. Informed consent was obtained from the parents and children before entering the study, which was approved by the local ethical committee (Institutional Review Board).

Patients will be randomly assigned in a double-blind manner to receive on the lesions 0.0003% calcitriol (Galderma, France), 0.1% tacrolimus (Astellas, Pharma, USA), and petrolatum (Aquaphor ointment)in all of them. All subjects were instructed to apply the treatment twice daily. Sunscreen will not be indicated, and hygienic habits are not being changed. Hypopigmented areas are going to be initially evaluated and supervised at 3, 6 and 9 weeks. Digital photographic registration(frontal, right, and left views) with an SLR Fuji FinepixS1pro camera will be taken and analysed by ImageJ software to quantify the reduction area of the plaques. The methods of assessment involve clinical evaluation by investigators, an independent observer, and by the transepidermal water loss (TEWL) with an evaporimeter (Dermalab, Cortex Technology, Denmark), and pigmentary changes using a colorimeter (Chromameter CR-300, Minolta, Osaka, Japan). Water loss will be recorded on each plaque for 60 seconds, as well as the L* (luminosity) and a* (erythema) axis. All adverse effects will be recorded. Statistical analysis was performed using T student, the level of significance was set at 5%. And clinical evaluation will be analysed by means of chi square tests.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Pityriasis alba with well defined lesions greater than 3 cm2.

Exclusion Criteria:

* Diagnosis of Atopic Dermatitis
* Skin disorders other than Pityriasis alba
* Systemic disorders
* Treatment during the last 8 weeks for this condition

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2008-01; Primary Completion 2010-08 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Repigmentation of PA lesions measured by colorimetry | 9 weeks
  Quantification of the repigmentation of lesions by means of the L axis of the CIE system. 0 is pure white, 100 y total dark.

SECONDARY OUTCOMES:
Change in transepidermal water loss of PA lesions | 6 weeks
  Quantification of water loss measured by a evaporimeter in grams per squared meter per hour. Is an indirect measure of stratum corneum integrity.
Investigator's repigmentation improvement | 9 weeks
  Clinical improvement is assessed by means of digital photographic registration (frontal, right, and left views). An independent observer clinically graded the global improvement as poor (0-25%), mild (26-50%), good (51-75%), and excellent (>75%).
Reduction of the affected area by image analysis software | 9 weeks
  ImageJ software will be used to measure the lesion reduction area after treatments

CONTACTS AND LOCATIONS:
Overall Officials: Juan P Castanedo-Cazares, MD, Study Chair — Dermatology Department. Hospital Central "Dr. Ignacio Morones Prieto". San Luis Potosi, México
Locations (1):
- Dermatology Department. Hospital Central "Dr. Ignacio Morones Prieto", San Luis Potosí City, San Luis Potosí, Mexico